CLINICAL TRIAL: NCT02057055
Title: The Effect of Surfactants on the Bacterial Composition of the Layers of the Skin
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: study not executed
Sponsor: University of California, San Diego (Other)
Responsible Party: Principal Investigator, Tissa Hata, MD, Clinical Professor of Medicine, University of California, San Diego
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: UCSD 131420
Record Dates: First submitted 2014-02-04; First posted 2014-02-06 (Estimated); Last update posted 2018-08-22 (Actual); Status verified 2018-08

CONDITIONS: Focus: Healthy Skin Microbiome
Keywords: Antibacterial soaps; Microbiome; Commensal bacteria; Pyrosequencing; Innate immunity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Soap 300000027003 (Experimental): Subjects will apply this soap to one of their arms daily in the shower for 3 weeks
  Interventions: Other: Soap 300000027003
- Soap 300000029240 (Experimental): Subjects will apply this soap to one of their arms daily in the shower for 3 weeks
  Interventions: Other: Soap 300000029240

INTERVENTIONS:
Other: Soap 300000027003
  Arms: Soap 300000027003
Other: Soap 300000029240
  Arms: Soap 300000029240

SUMMARY:
Recent research in the investigator's lab has shown that bacteria are present not only on the outer surface of our skin, but also in the deeper components as well. In this study, the investigator will study the bacteria present in different components of the skin including the epidermis, dermis, subcutaneous fat, and hair follicle, and determine if and how these bacteria change after repeated use of different commercially available hand soaps. It is expected that the bacteria populations in the different skin components will change with the use of different soaps.

DETAILED DESCRIPTION:
This study will consist of 5 visits over approximately 2 months. All study procedures will occur at the University of California San Diego Division of Dermatology Outpatient Clinic. The procedures for each visit will be described below.

Visit 1 (Day 0) At this visit, after obtaining informed consent from subjects, the inclusion/exclusion criteria will be reviewed. This step will require a brief medical history and skin examination to be performed. Both the history and physical exam will be performed by a licensed physician. Eligible subjects will proceed with the remainder of the study. These subjects will be provided with a mild soap (ID# 100000049586) to use whenever they shower for the remainder of the study. These subjects will also be instructed that they may not apply any topical lotions, creams, or other products to their arms during the remainder of the study. Subjects will also be told to avoid excessive sun exposure on their arms, including tanning or the use of tanning beds, while participating in this study.

Visit 2 (Day 14) Subjects will return on Day 14 for Visit 2. Any adverse events will be recorded, and the subject's interim medical history will be taken. Two skin swabs will then be taken from the skin on subject's the upper inner arm. One swab will be from the right arm and the other from the left arm. A 4-mm punch biopsy will then be taken from one of the arms near the area that was swabbed. To perform this procedure, the skin is injected with about 1-2 cc of local anesthetic. A 4 mm punch will be used to remove the biopsy specimen from the location previously agreed upon by the investigator and subject. A 4.0 nylon suture will be used to close the biopsy site, and ointment and a Band-Aid applied.

Visit 3 (Day 28 +/- 4) Subjects will return around Day 28 for their third visit. At this visit, any adverse events since the last visit will be recorded, and the subject's interim medical history will be taken. The suture will be removed from the site of the biopsy taken at Visit 2. Subjects will then be provided with two body washes (ID# 300000027003 and ID# 300000029240) to use in the shower when washing their upper inner arms. One soap will be used to wash the upper half of the right arm, and the other soap will be used to wash the upper half of the left arm. The subject will continue using the Mild Body Wash in the shower when washing all other body parts. The subject will also be instructed not to apply any other creams, ointments or medications to their arms, and to avoid excess sun exposure to their upper arms during this time.

Visit 4 (Day 49 +/- 4) Subjects will return around Day 49 for their next visit. Any adverse events as well as changes to their interim medical history since their last visit will be recorded. A skin swab of each upper inner arm will then be taken. A 4-mm punch biopsy will then be taken from an area of skin in the upper inner region of both the right and left arms for a total of 2 biopsies taken during this visit. At the termination of this visit, subjects can resume use of their normal shower production and application of any creams or lotions they normally use on their arms.

Visit 5 (Day 59 +/- 4) Subjects will return on this day to have their sutures removed. Any adverse events will be recorded. This visit will conclude all study-related activities.

All samples will be processed in the lab. Skin swabs will undergo pyrosequencing to determine the different strains of bacteria present on the subject's skin, as well as quantitative polymerase chain reaction to determine the abundance of S. aureus, S. epidermidis, and P. acnes on each subject's skin surface. Biopsy specimens will be sectioned and each section will be placed on a glass slide. The sections will undergo immunostaining to stain for bacteria. Laser-capture microdissection of each section into its four skin components will be used to assist in evaluating the bacteria present in the different skin layers.

ELIGIBILITY:
Inclusion Criteria:

* Age 21-35 years
* Male subject of any race and ethnicity
* Subject agrees to comply with study requirements

Exclusion Criteria:

* Subjects with severe medical condition(s) that in the view of the investigator prohibits participation in the study
* Dermatologic disease such as psoriasis or atopic dermatitis which may have inherently abnormal antimicrobial peptide levels
* Subject has Netherton's syndrome or other genodermatoses that result in a defective epidermal barrier
* Pregnant or nursing females
* Immunocompromised subjects (e.g., lymphoma, HIV/AIDS, Wiskott-Aldrich Syndrome), or with a history of active or malignant disease (excluding non-melanoma skin cancer) as determined by the participant's medical history.
* Subjects with a history of psychiatric disease or history of alcohol or drug abuse that would interfere with the ability to comply with the study protocol
* Active viral or fungal skin infections at the target areas
* Are currently receiving lithium, antimalarials, or intramuscular gold now or within the last 4 weeks.
* Ongoing participation in an investigational drug trial
* Use of any oral or topical antibiotic during the study and up to one week prior to entering the study
* Use of any local topical medications less than one week prior to screening
* Use of any systemic immunosuppressive therapy less than four weeks prior to screening.
* Subjects with a history of or propensity to developing reactions after use of over the counter cleansers
* Subjects with diabetes
* Injured, broken skin
* Allergy to local anesthetic medications, including lidocaine

Ages: 21 Years to 35 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 0 (Actual)
Dates: Start 2014-02; Primary Completion 2016-08 (Estimated); Study Completion 2016-08 (Estimated)

PRIMARY OUTCOMES:
Number of bacteria | 3 weeks
  The number of bacteria present on/in the epidermis, dermis, subcutaneous fat and hair follicle will be determined using both polymerase chain reaction and colony counting methods after subjects have used each of the body washes on their arms for a total of 3 weeks.

SECONDARY OUTCOMES:
Type of bacteria | 3 weeks
  The type (i.e. strain) of bacteria present on the skin surface will be determined after subjects use each of the body washes on their arms for three weeks
Change in type of bacteria | 3 weeks
  The change in the type (i.e. strain) of bacteria present on the skin surface will be determined after subjects use each of the body washes on their arms for three weeks and compared to the types of bacteria present at the time of the baseline swabs
Change in number of bacteria | 3 weeks
  The change in the number of bacteria present in the different skin compartments will be determined after subjects use each of the body washes on their arms for three weeks and compared to the number of bacteria present at the time of the baseline biopsies
Type of bacteria | Baseline
  The baseline type (i.e. strain) of bacteria present on the skin surface will be determined after subjects use a mild body wash on their arms for two weeks
Number of bacteria | Baseline
  The baseline number of bacteria present on the skin surface will be determined after subjects use each a mild body wash for two weeks

CONTACTS AND LOCATIONS:
Overall Officials: Tissa Hata, MD, Principal Investigator — University of California, San Diego
Locations (1):
- University of California San Diego Division of Dermatology, San Diego, California, United States